CLINICAL TRIAL: NCT00494533
Title: Treprostinil for Untreated Symptomatic PAH Trial: A 12-Week Multicenter Randomized Double-Blind Placebo-Controlled Trial of the Safety and Efficacy of Intravenous Remodulin® in Patients in India With Pulmonary Arterial Hypertension
Brief Title: Study of Intravenous Remodulin in Patients in India With Pulmonary Arterial Hypertension
Acronym: TRUST-1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Safety issues related to outpatient intravenous infusion in India
Sponsor: United Therapeutics (Industry)
Collaborators: Asian Clinical Trials (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIV-PH-402
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; prostacyclin analogue; intravenous
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Remodulin (treprostinil sodium)

SUMMARY:
Multi-center, double-blind, placebo-controlled, randomized, parallel study comparing continuous intravenous (IV) Remodulin® to placebo in patients with pulmonary arterial hypertension either primary (PPH) or associated with human immunodeficiency virus (HIV) infection or collagen vascular disease).

ELIGIBILITY:
Inclusion Criteria: Patients Must

1. Between 16- 75 years of age.
2. Male or, if female, physiologically incapable of childbearing or utilizing birth control.
3. Have current diagnosis of symptom-limited NYHA Functional Class III/IV PAH that is:

   * PPH ("idiopathic" or familial PAH); or
   * PAH associated with collagen vascular disease (confirmed by antinuclear antibody titer or acceptable test); or
   * PAH associated with HIV infection (confirmed by serological test).
4. If HIV positive, have CD4 lymphocyte count ≥ 200 at baseline and receiving current SOC anti-retroviral or effective medication for HIV infection.
5. Optimally treated with conventional PH therapy and clinically stable for at least 1 month prior to baseline.
6. Have ventilation/perfusion scan, contrast-enhanced CT scan, or pulmonary angiogram after onset of PAH that rules out pulmonary embolism.
7. Have cardiac catheterization in last 3 months (or at Baseline) showing:

   * PAPm > 35 mmHg (at rest) &
   * PCWPm (or LV end diastolic pressure) < 16 mmHg &
   * PVR > 5 mmHg/L/min.
8. Have echocardiogram in last 3 months consistent with PH, specifically:

   * evidence of RV hypertrophy or dilation &
   * evidence of normal LV function &
   * absence of mitral valve stenosis.
9. Have chest radiograph consistent with PH performed in last 3 months. Radiograph must show clear lung fields or no more than patchy interstitial infiltrates.
10. Unless contraindicated, able to receive one of following anticoagulants: warfarin to achieve INR between 1.5-2.5 or heparin to produce aPTT between 1.3-1.5 times control, unless higher levels clinically indicated.
11. Mentally and physically capable of learning to administer Study Drug using ambulatory intravenous infusion pump and central venous access, or have trained caregiver.
12. If on corticosteroids, receiving stable dose of 20 mg/day of prednisone (or equivalent dose of another steroid) for at least 1 month prior to entry.

Exclusion Criteria: Patients must not:

1. Nursing or pregnant (women of childbearing potential have negative pregnancy test).
2. Have had new type of chronic therapy (including but not limited to oxygen, different category of vasodilator, diuretic, digoxin) for PH, except for anticoagulants, added in last month.
3. Be scheduled for heart-lung transplant.
4. Have any PH medication except for anticoagulants discontinued in week prior to study entry.
5. Have received any chronic prostaglandin or prostaglandin analogue (including intravenous/inhaled/oral: epoprostenol, iloprost, beraprost, etc.), any phosphodiesterase inhibitor therapy such as sildenafil, or any endothelin antagonist therapy such as bosentan, in past 30 days.
6. Have PH associated with chronic thromboembolic disease; or chronic obstructive lung diseases or hypoxemia; or evidence of significant parenchymal lung disease as evidenced by PFTs in last 3 months as follows (any one of following):

   * TLC < 60% (predicted) or high resolution CT documenting diffuse interstitial fibrosis or alveolitis
   * FEV1/FVC ratio < 50%
7. Have Portal Hypertension.
8. Have history of uncontrolled Sleep Apnea, defined as oxygen desaturation less than 90% at night, in past 3 months.
9. Have history of left-sided heart disease including:

   * Aortic or mitral valve disease or
   * Pericardial constriction or
   * Restrictive or congestive cardiomyopathy; or have evidence of current left-sided heart disease defined by:
   * PCWPm or LV end diastolic pressure > 16 mmHg or
   * LVEF < 40% by MUGA, angiography or echocardiography or
   * LV Shortening Fraction < 22% by echocardiography or
   * Symptomatic coronary disease (demonstrable ischemia).
10. Have any disease other than HIV or connective tissue disease associated with PH (e.g. sickle cell anemia, schistosomiasis).
11. Have active AIDS or tuberculosis.
12. Have musculoskeletal disorder (e.g. arthritis, artificial leg, etc.) or any other disease thought to limit ambulation, or connected to machine which is not portable.
13. Have baseline exercise capacity of <50 m or >325 m as measured by 6-Minute Walk Test.
14. Have uncontrolled systemic hypertension as evidenced by systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg.
15. Have used prescription appetite suppressants in 3 months of study entry.
16. Have chronic renal insufficiency defined by creatinine >2.5 mg/dL or requiring dialysis.
17. Receiving an investigational drug (other than acute challenge with epoprostenol), have in place an investigational device, or have participated in investigational drug/device study in past 30 days.
18. Have presence of any physiological or mental condition which contraindicates administration of Remodulin.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Six-minute walk distance | Twelve Weeks
  Placebo-corrected change in 6-minute walk distance from Baseline to Week 12.

SECONDARY OUTCOMES:
Borg Dyspnea Score | Twelve Weeks
  The Bord dyspnea score is a 10-point scale rating the maximum level of dyspnea experienced during the six-minute walk test (6MWT). The Borg dyspnea score was assessed immediately following the 6MWT. Scores ranged from 0 (for no shortness of breath) to 10 (for greatest shortness of breath ever experienced).
Dyspnea-Fatigue Index | Twelve weeks
  The dyspnea-fatigue index was assessed at Baseline, Weeks 1, 4, 8 ans 12. Each of the three components of the dyspnea-fatigue index were rated on a scale of 0 to 4, with 0 being the worst condition and 4 being the best condition for each component. The dyspnea-fatigue index is computed by summing the three component scores.
NYHA Functional Class | Twelve Weeks
  Changes from Baseline in NYHA Functional Class will be summarized and compared between treatment groups at Weeks 1, 4, 8 and 12.
Clinical Worsening | Twelve Weeks
  Clinical worsening was defined as worsening PAH resulting in death, transplant, hospitalization, necessity to unblind for rescue therapy, or an inability to physically perform the walk assessment. Incidence of clinical worsening and the time from Baseline to clinical worsening will be compared between treatment groups.
Combined Walk and Borg Dyspnea Score | 12 Weeks
  The intent of the Six-Minute Walk Test is to determine how much patients can do during the course of carrying out activities of daily living. However, the capacity of patients to function is determined not only by what they can do when they exert themselves to the fullest, but also by how they feel when they are carrying out their usual activities of daily living. It is therefore important not only to look at the distance traversed during the unencouraged 6-minute walk but also the symptoms experienced at the end of the effort. To do so, walk distances and Borg Scores from the Week 12 Six-Minute Walk Test were simultaneously compared between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wade, Ph.D., Study Director — United Therapeutics
Locations (14):
- India (14):
  - SAL Hospital & Medical Institute, Ahmedabad
  - Narayana Hrudayalaya Inst. Of Cardiac Sciences, Bangalore
  - Apollo Hospitals, Chennai
  - K. S. Hospital, Chennai
  - Sri Ramachandra Medical College, Chennai
  - Medwin Heart Institute, Hyderabad
  - Yashoda Super Specialty Hospital, Hyderabad
  - Apollo Gleneagles Hospital, Kolkata
  - KMC Hospital, Mangalore
  - Kasturba Medical College, Manipal
  - KEM Hospital, Mumbai
  - G. B. Pant Hospital & Maulana Azad Med. College, New Delhi
  - Ruby Hall Clinic, Pune
  - Krishna Institute of Medical Sciences, Secunderabad

REFERENCES:
- [Derived] Hiremath J, Thanikachalam S, Parikh K, Shanmugasundaram S, Bangera S, Shapiro L, Pott GB, Vnencak-Jones CL, Arneson C, Wade M, White RJ; TRUST Study Group. Exercise improvement and plasma biomarker changes with intravenous treprostinil therapy for pulmonary arterial hypertension: a placebo-controlled trial. J Heart Lung Transplant. 2010 Feb;29(2):137-49. doi: 10.1016/j.healun.2009.09.005. PMID 20022264